CLINICAL TRIAL: NCT01119911
Title: Blood Sampling Through Peripheral Venous Catheter for Selected Basic Analytes in Infants
Brief Title: Blood Sampling Through Peripheral Venous Catheter in Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10086-09CTIL
Record Dates: First submitted 2010-05-04; First posted 2010-05-10 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Pain
Keywords: Blood sampling; Venipuncture; Peripheral venous catheter; Complete blood count; Basic chemistry; Hemolysis; Peripheral venous catheter replaces venipuncture.; Peripheral venous catheter blood sampling reduces pain.
MeSH Terms: conditions — Pain; Hemolysis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sampling from peripheral venous catheter. — Venipuncture is performed on the opposite limb of the peripheral venous catheter. Within 3 minutes, a second sample is taken from existing peripheral venous catheter used for fluid administration. Intravenous fluids are then stopped for 30 seconds and a tourniquet applied proximal to the device for another 30 seconds. A 2-mL syringe is attached and 0.5 mL of blood aspirated and discarded. Thereafter, 2 mL blood is slowly drawn during about 15 seconds, into a different 2-mL syringe, to allow a gentle pumping action that may reduce vacuum in the syringe and thus hemolysis rates. Afterwards, the intravenous device is flushed with 2 mL normal saline and infusion restarted.

SUMMARY:
We hypothesize that peripheral venous catheter used for fluid administration can replace venipuncture blood sampling for selected basic analytes and thus reduce pain in infants under 2 years of age.

DETAILED DESCRIPTION:
Multiple venipunctures in hospitalized children result in physical and emotional distress. Recently, we have found that blood sampling via peripheral venous catheter used for fluid administration in children significantly reduces pain and, except for glucose, can replace venipuncture for determining complete blood count and basic chemistry analytics, including white and red blood cell counts, hemoglobin and hematocrit levels, mean corpuscular volume, mean corpuscular hemoglobin level, red blood cell distribution width, platelet count, mean platelet volume, and sodium, potassium, chloride, and urea levels (Berger-Achituv S, Budde-Schwartzman B. Ellis MH, Shenkman Z. Erez I. Blood Sampling through Peripheral Venous Catheters for Selected Basic Analytes in Children. Pediatrics. In press).

The goal of this study is to investigate whether blood sampling via peripheral venous catheter used for fluid administration can significantly reduces pain and replace venipuncture for determining complete blood count and basic chemistry analytics in infants under 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 2 years of age.
* Only hemodynamically stable infants.
* Infants with peripheral venous catheter present for less than 72 hours.
* At least 20 mL of fluids have been infused intravenously at the time of blood sampling.

Exclusion Criteria:

* Infants with signs of catheter-related thrombophlebitis.

Ages: 1 Week to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants under 2 years of age, admitted to the Departments of Pediatrics and Pediatric Surgery, Meir Medical Center, who have a functioning peripheral venous catheter and require repeated blood sampling for diagnostic purposes.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the interchangeability of peripheral venous catheter and venipuncture for complete blood count and basic chemistry indices. | Primary assessment will be done after data analysis of the first 20 participants, estimated to take up to 3 months.
  Comparisons of complete blood count (including white and red blood cells, hemoglobin, hematocrit, mean corpuscular volume and hemoglobin, red cell distribution width, platelets, mean platelet volume) and basic chemistry indices (including sodium, potassium, glucose, chloride, urea) will be performed and hemolysis will be documented.

SECONDARY OUTCOMES:
Assessment of infant's mood during procedures. | Primary assessment will be done after data analysis of the first 20 participants, estimated to take up to 3 months.
  The investigator will record infant's mood (calm, distressed/crying, crying vigorously) during blood sampling from peripheral venous catheter and direct venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Sivan Berger-Achituv, MD, Principal Investigator — Meir Medical Center; Ilan Erez, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel